CLINICAL TRIAL: NCT04662203
Title: Is Frailty a Prognostic Factor for Relevant Outcomes in the Management of Hypertension in Older People, and is There Evidence That the Association of Blood Pressure and Outcomes is Different in the Context of Frailty?
Brief Title: Can Frailty Inform the Management of Hypertension in Older People?
Acronym: Frail_BP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leeds (Other)
Collaborators: Swansea University (Other); University of Oxford (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Oliver Todd, Dunhill Medical Trust doctoral research fellow, University of Leeds
Other Study IDs: RTF107/0117
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Hypertension; Frailty
MeSH Terms: conditions — Hypertension; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to investigate in large scale routine primary care data whether frailty is a prognostic factor for relevant outcomes in the management of hypertension in older people and whether frailty causes effect modification of the association of blood pressure or blood pressure lowering treatment and outcomes in older people.

DETAILED DESCRIPTION:
A retrospective cohort study used linked electronic health records from the Welsh Secure Anonymised Information Linkage (SAIL) databank. All patients had hypertension in the absence of established cardiovascular disease, and were over the age of 65 years in 2007. Systolic blood pressure and frailty, measured using the electronic frailty index were recorded. Patients were followed up for ten years. Time to event analysis measured first ever major adverse cardiovascular or cerebrovascular event (MACCE), all-cause mortality and injurious falls. Adjustment was made for established cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient registered with a general practitioner contributing to SAIL database for at least 1 year
* Patient with blood pressure measured and recorded at any time after 1st January 2007 and before 1st January 2008, was used as the individual's index start date.
* Patient aged 65 years or older at the time of study entry.

Exclusion Criteria:

* Patient did not have a diagnosis of hypertension or did not have blood pressure meeting criteria for hypertension;
* Patient had an established history of cardiovascular disease (previous stroke, heart failure or myocardial infarction) prior to the start date.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients living in the community registered with a general practitioner in Wales.
Sampling Method: Non-Probability Sample
Enrollment: 145598 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | 10 years
  Myocardial infarction; stroke; new diagnosis of heart failure; cardiovascular death

SECONDARY OUTCOMES:
All-cause mortality | 10 years
  Death from any cause
Injurious falls | 10 years
  Fall leading to fracture of bone and hospital admission

IPD SHARING:
Plan to Share IPD: Undecided